CLINICAL TRIAL: NCT03337867
Title: Theta-Burst-Stimulation in Recurrent Stroke Recovery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Christian Grefkes, Principal Investigator, Professor, University Hospital of Cologne
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: U1111-1204-6783
Record Dates: First submitted 2017-11-03; First posted 2017-11-09 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Stroke; Neurorehabilitation
Keywords: Recurrent stroke; Stroke; Transcranial Magnetic Stimulation; Theta-Burst-Stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-iTBS (Active Comparator)
  Interventions: Device: Magstim Super Rapid2 System
- Sham-iTBS (Sham Comparator)
  Interventions: Device: Magstim Super Rapid2 System

INTERVENTIONS:
Device: Magstim Super Rapid2 System — Intermittent theta-burst-stimulation (iTBS) protocol
  Arms: Real-iTBS
Device: Magstim Super Rapid2 System — Sham stimulation
  Arms: Sham-iTBS

SUMMARY:
The present study aims at investigating the effects of intermittent theta-burst stimulation (iTBS) for motor recovery in recurrent stroke patients. Therefore a daily intervention of repetitive transcranial magnetic stimulation over 8 days combined with subsequent physiotherapy is compared to a control condition, sham stimulation combined with subsequent physiotherapy. Motor function, degree of disability and quality of life are examined in order to evaluate the effects of iTBS in the rehabilitation of recurrent stroke patients in the first weeks and after three months.

DETAILED DESCRIPTION:
To date, the majority of neuromodulation approaches aiming at improving motor recovery after stroke are limited to patients with first-ever ischemic stroke. Therefore, rehabilitation of recurrent stroke mainly includes physiotherapy and occupational therapy. Yet, particular these patients retain movement impairment relevant for activities of daily living.

By using repetitive transcranial magnetic stimulation (rTMS), it is possible to promote recovery of connectivity between brain regions, particularly after stroke and thereby improve motor performance. Previous data indicate that intermittent theta-burst stimulation (iTBS), a protocol of neuromodulation, enhances the effects of subsequent motor training in early rehabilitation after stroke.

The current study aims at investigating whether daily repetitive transcranial magnetic stimulation over 8 days combined with subsequent physiotherapy leads to better motor recovery in recurrent stroke, compared to control condition, physiotherapy after sham stimulation. Motor function, degree of disability and quality of life are examined in order to evaluate the effects of iTBS in the rehabilitation of recurrent stroke patients in the first weeks and after three months.

ELIGIBILITY:
Inclusion Criteria:

* written consent
* age: 40-90 years
* recurrent stroke
* hemiparesis with impaired hand motor function

Exclusion Criteria:

* Subjects who are legally detained in an official institute (§20 MPG)
* Electronic implants or ferromagnetic Implants located in the head, neck or thorax (e.g. clips, intracranial shunt, artificial heart valve, pacemaker)
* Medication pump (e.g. insulin pump)
* Metal splinters in eye or head
* Pregnancy / breastfeeding
* Severe Neurodegenerative disease
* Severe Neuroinflammatory disease
* History of seizures / epilepsy
* Physical addiction to alcohol, medication, or drugs (excluded: nicotine)
* Insufficient compliance
* Present or past malignant tumor involving the central nervous system
* Severe Psychiatric disease
* Frequent medication with benzodiazepines, high-potency antipsychotics or tricyclic antidepressants before hospitalization or long-term during hospitalization

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-11 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Relative grip force | 3 months after enrollment
  grip force as measured with vigorimeter

SECONDARY OUTCOMES:
Relative grip force | After 8 days of intervention, and 3 months of enrollment
  Grip force as measured with vigorimeter
Motor function | After 8 days of intervention, and 3 months of enrollment
  Action Research Arm Test, ARAT
Motor function | After 8 days of intervention, and 3 months of enrollment
  Fugl-Meyer Motor Scale of the upper extremity, FM The Fugl-Meyer Assessment scale is an ordinal scale that has 3 points for each item. A zero score is given for the item if the subject cannot do the task. A score of 1 is given when the task is performed partially and a score of 2 is given when the task is performed fully.
  Minimum score in upper limb = 0 Maximum score in upper limb = 66, Subscales are summed
Stroke severity | After 8 days of intervention, and 3 months of enrollment
  National Instituts of Health Stroke Scale, NIHSS The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.
  The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Degree of disability | After 8 days of intervention, and 3 months of enrollment
  Modified Rankin Scale, mRS The scale runs from 0-6, running from perfect health (0) without symptoms to death (6).
Motor cortex excitability/ Motor evoked potential | After 8 days of intervention, and 3 months of enrollment
  Motor evoked potential (MEP) induced by stimulation of the affected motor cortex
Motor cortex excitability/ Resting motor threshold | After 8 days of intervention, and 3 months of enrollment
  Resting motor threshold as measured by stimulation of the affected motor cortex, RMT
Motor cortex excitability/ Short-interval intracortical inhibition | After 8 days of intervention, and 3 months of enrollment
  Short-interval intracortical inhibition Short-interval intracortical inhibition (SICI) is a widely used paired-pulse transcranial magnetic stimulation (TMS) measure to assess inhibition in human motor cortex
Motor cortex excitability/ Ipsilateral silent period | After 8 days of intervention, and 3 months of enrollment
  Ipsilateral silent period The ipsilateral silent period (iSP) is supposed to be a specific marker of transcallosal motor inhibition. Measured by a short attenuation or interruption of ongoing voluntary electromyographic (EMG) activity in hand muscles induced by focal TMS of the ipsilateral M1.
Quality of life | After 8 days of intervention, and 3 months of enrollment
  EuroQol 5D questionnaire, EQ-5D
Activities of daily living at admission and discharge in external rehabilitation facility | After 8 days of intervention, and 3 months of enrollment
  Barthel-Index (BI) scores as documented by external rehabilitation facility The Barthel scale is an ordinal scale used to measure performance in activities of daily living (ADL). A higher number is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital. The scale yield a score of 0-100.
Days of rehabilitation after intervention phase | 3 months after enrollment
  Days of rehabilitation after intervention phase as documented by external rehabilitation facility

CONTACTS AND LOCATIONS:
Overall Officials: Christian Grefkes, MD, Principal Investigator — University Hospital Cologne
Locations (1):
- Christian Grefkles, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No